CLINICAL TRIAL: NCT00560053
Title: Multiple Myeloma 2000. Multicentric Evaluation of a Therapeutic Strategy Optimized in Multiple Myeloma. Analysis of Efficiency and Possible Pronostic Impact of Minimal Residual Disease (Measured By PCR And Citometry of Flow) in Patients With Complete Response
Brief Title: Pethema Multiple Myeloma 2000
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA MM-2000
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Alternating chemotherapy; Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Transplantation, Autologous; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alternating chemotherapy — 4 cycles of alternating chemotherapy VBMCP/VBAD (every 5 weeks). VBMCP: Vcr 2 mg ev day 1, BCNU 0.5 mg/kg ev day 1, Cyclophosphamide 10 mg/kg day 1, Melphalan 0.25 mg/kg v.o. days 1-4, Prednisone 1 mg/kg v.o. days 1-4, 0.5 mg/kg days 5-8 and 0.25 mg/kg days 9-12.
  VBAD: Vcr 1 mg e.v. day 1, BCNU 30 mg/m 2 e.v. day 1, Adriamycine 40 mg/m 2 day 1, Dexamethasone 40 mg/m 2 days 1-4, 9-12 and 17-20.
Procedure: Autologous Transplantation — Autologous Transplantation :
  BUMEL:Busulfan, total dose 12 mg/kg (days -6 a -3; prophylaxis with difenilhidantoine) Melphalan 140 mg/m 2 , ev day -2 TASPE: To investigator criteria
Drug: Maintenance — At 3 months of transplantation or with >1.500 neutrophiles/ > 75.000 platelets mm 3 .
  Prednisone: 50 mg alternating days during 2 years Interferon alfa 2-b: 3 M UI s.c. Three times a week until relapse.
Procedure: Second transplantation — In cases that no reach CR with BUMEL is programmed second transplantation, after 4-8 months .
Procedure: ALOGENIC MINI TRASPLANTATION — ALOGENIC MINI TRASPLANTATION Fludarabine 30 mg / m 2 / day, days -7, -6, -5, -4, -3 Melphalan 70 mg / m 2 / day, day -2 Prophylaxis EICH: CsA + MTX or CsA + MOFETIL

SUMMARY:
The study objectives are to investigate the toxicity and the BUMEL response rate; in patients who reach the CR after autotransplantation, investigate if negativization of IF, influences in disease evolution; in patients in PR after autotransplantation, analyze if the second intensive procedure is capable of increasing the response rate and increasing the survival so that patients who reached the CR with the first transplantation; Patients with MM primarily resistant to the chemotherapy, investigate the efficacy of a double transplantation; patients submitted to double transplantation, control the efficacy of the second transplantation in front of allogenic transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Less 70 years
* ECOG 0-2
* Symptomatic MM (pain, anemia, infection, haemorrhage, loss of weight, hypercalcemia, extramedulary plasmocytoma, creatinine >2 mg/dl).
* No previous chemotherapy

Exclusion Criteria:

* >70 years
* ECOG 3-4
* myeloma quiescent
* cardiopathy
* liver disfunction
* HIV+
* Hepatitis B-C +
* Previous chemotherapy

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2000-01; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bladé, Dr, Study Chair — Hospital Clinic of Barcelona; Juan Jose Lahuerta, Dr, Study Chair — Hospital Doce de Octubre Madrid; Adrián Alegre, Dr, Study Chair — Hospital La Princesa Madrid; Anna Sureda, Dr, Study Chair — Hospital Sant Pau Barcelona; Joaquín Díaz Mediavilla, Dr, Study Chair — Hospital Clinico Madrid; Javier De la Rubia, Dr, Study Chair — Hospital La Fe de Valencia; Joan Bargay, Dr, Study Chair — Hospital Son Dureta Palma de Mallorca; Jose García-Laraña, Dr, Study Chair — Hospital Universitario Ramon y Cajal; Eulogio Conde, Dr, Study Chair — Hospital Valdecilla Santander; Felipe Prosper, Dr, Study Chair — Hospital Clinico Valencia

REFERENCES:
- [Derived] Martinez-Lopez J, Fernandez-Redondo E, Garcia-Sanz R, Montalban MA, Martinez-Sanchez P, Pavia B, Mateos MV, Rosinol L, Martin M, Ayala R, Martinez R, Blanchard MJ, Alegre A, Besalduch J, Bargay J, Hernandez MT, Sarasquete ME, Sanchez-Godoy P, Fernandez M, Blade J, San Miguel JF, Lahuerta JJ; GEM (Grupo Espanol Multidisciplinar de Melanoma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) cooperative study group. Clinical applicability and prognostic significance of molecular response assessed by fluorescent-PCR of immunoglobulin genes in multiple myeloma. Results from a GEM/PETHEMA study. Br J Haematol. 2013 Dec;163(5):581-9. doi: 10.1111/bjh.12576. Epub 2013 Oct 3. PMID 24117042
- [Derived] Blanes M, Lahuerta JJ, Gonzalez JD, Ribas P, Solano C, Alegre A, Blade J, San Miguel JF, Sanz MA, de la Rubia J. Intravenous busulfan and melphalan as a conditioning regimen for autologous stem cell transplantation in patients with newly diagnosed multiple myeloma: a matched comparison to a melphalan-only approach. Biol Blood Marrow Transplant. 2013 Jan;19(1):69-74. doi: 10.1016/j.bbmt.2012.08.009. Epub 2012 Aug 13. PMID 22897964
- [Derived] Rosinol L, Garcia-Sanz R, Lahuerta JJ, Hernandez-Garcia M, Granell M, de la Rubia J, Oriol A, Hernandez-Ruiz B, Rayon C, Navarro I, Garcia-Ruiz JC, Besalduch J, Gardella S, Lopez Jimenez J, Diaz-Mediavilla J, Alegre A, San Miguel J, Blade J; PETHEMA/Spanish Myeloma Group. Benefit from autologous stem cell transplantation in primary refractory myeloma? Different outcomes in progressive versus stable disease. Haematologica. 2012 Apr;97(4):616-21. doi: 10.3324/haematol.2011.051441. Epub 2011 Nov 4. PMID 22058223
- [Derived] Lahuerta JJ, Mateos MV, Martinez-Lopez J, Grande C, de la Rubia J, Rosinol L, Sureda A, Garcia-Larana J, Diaz-Mediavilla J, Hernandez-Garcia MT, Carrera D, Besalduch J, de Arriba F, Oriol A, Escoda L, Garcia-Frade J, Rivas-Gonzalez C, Alegre A, Blade J, San Miguel JF; Grupo Espanol de MM and Programa para el Estudio de la Terapeutica en Hemopatia Maligna Cooperative Study Groups. Busulfan 12 mg/kg plus melphalan 140 mg/m2 versus melphalan 200 mg/m2 as conditioning regimens for autologous transplantation in newly diagnosed multiple myeloma patients included in the PETHEMA/GEM2000 study. Haematologica. 2010 Nov;95(11):1913-20. doi: 10.3324/haematol.2010.028027. Epub 2010 Jul 27. PMID 20663944
- [Derived] Paiva B, Vidriales MB, Perez JJ, Mateo G, Montalban MA, Mateos MV, Blade J, Lahuerta JJ, Orfao A, San Miguel JF; GEM (Grupo Espanol de MM) cooperative study group; PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) cooperative study group. Multiparameter flow cytometry quantification of bone marrow plasma cells at diagnosis provides more prognostic information than morphological assessment in myeloma patients. Haematologica. 2009 Nov;94(11):1599-602. doi: 10.3324/haematol.2009.009100. PMID 19880781
- [Derived] Paiva B, Vidriales MB, Mateo G, Perez JJ, Montalban MA, Sureda A, Montejano L, Gutierrez NC, Garcia de Coca A, de las Heras N, Mateos MV, Lopez-Berges MC, Garcia-Boyero R, Galende J, Hernandez J, Palomera L, Carrera D, Martinez R, de la Rubia J, Martin A, Gonzalez Y, Blade J, Lahuerta JJ, Orfao A, San-Miguel JF; GEM (Grupo Espanol de MM)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Groups. The persistence of immunophenotypically normal residual bone marrow plasma cells at diagnosis identifies a good prognostic subgroup of symptomatic multiple myeloma patients. Blood. 2009 Nov 12;114(20):4369-72. doi: 10.1182/blood-2009-05-221689. Epub 2009 Sep 15. PMID 19755674
- [Derived] Paiva B, Vidriales MB, Cervero J, Mateo G, Perez JJ, Montalban MA, Sureda A, Montejano L, Gutierrez NC, Garcia de Coca A, de Las Heras N, Mateos MV, Lopez-Berges MC, Garcia-Boyero R, Galende J, Hernandez J, Palomera L, Carrera D, Martinez R, de la Rubia J, Martin A, Blade J, Lahuerta JJ, Orfao A, San Miguel JF; GEM (Grupo Espanol de MM)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Groups. Multiparameter flow cytometric remission is the most relevant prognostic factor for multiple myeloma patients who undergo autologous stem cell transplantation. Blood. 2008 Nov 15;112(10):4017-23. doi: 10.1182/blood-2008-05-159624. Epub 2008 Jul 31. PMID 18669875
- [Derived] Rosinol L, Perez-Simon JA, Sureda A, de la Rubia J, de Arriba F, Lahuerta JJ, Gonzalez JD, Diaz-Mediavilla J, Hernandez B, Garcia-Frade J, Carrera D, Leon A, Hernandez M, Abellan PF, Bergua JM, San Miguel J, Blade J; Programa para el Estudio y la Terapeutica de las Hemopatias Malignas y Grupo Espanol de Mieloma (PETHEMA/GEM). A prospective PETHEMA study of tandem autologous transplantation versus autograft followed by reduced-intensity conditioning allogeneic transplantation in newly diagnosed multiple myeloma. Blood. 2008 Nov 1;112(9):3591-3. doi: 10.1182/blood-2008-02-141598. Epub 2008 Jul 8. PMID 18612103
- See also: spanish hematology association — http://aehh.org